CLINICAL TRIAL: NCT03626025
Title: Randomized Prospective Study Comparing the Effectiveness of Massed and Spaced Learning in Microsurgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hand & Reconstructive Microsurgery (Other)
Responsible Party: Sponsor-Investigator, Hand & Reconstructive Microsurgery, Head of Department, Dr Alphonsus Khin Sze Chong, National University Hospital, Singapore
Organization: National University Hospital, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016/01133
Record Dates: First submitted 2018-06-24; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Mass Learning, Spaced Learning, Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mass Learning Group (No Intervention): Participants underwent an eight-hour microsurgery training course in a single session under the mass-learning format.
- Spaced Learning Group (Other): Participants underwent two-hour microsurgery training sessions every week for a total of 4 sessions under the spaced learning format.
  Interventions: Other: Spaced learning

INTERVENTIONS:
Other: Spaced learning — Instead of learning over a single session, teaching is carried out over a few weekly sessions but maintaining the overall total number of hours spent on teaching
  Arms: Spaced Learning Group

SUMMARY:
Title: Randomized prospective study comparing the effectiveness of spaced learning to mass learning in microsurgical procedures.

Background:

Spacing phenomenon occurs when learning outcomes are greater with the teaching process spread out over time (spaced learning), as opposed to having the same total duration of teaching carried out over a single session (mass learning). Spaced learning has been shown to improve explicit memory tasks including free recall, recognition, cued -recall and frequency estimation. It has been used in various medical specialties with promising results and has been shown to be at least as good as mass training in learning clinical skills such as cardio-pulmonary resuscitation and laparoscopy skills.

We aim to test the concept of spaced learning in learning delicate and complex skilled procedures like microsurgery. Our hypothesis is that spaced learning is better than mass learning in acquiring microsurgical suturing skills.

Methodology:

Medical students with no prior exposure to microsurgical training were randomized into control (mass-learning) and treatment (spaced learning) groups. The students were all taught to handle microsurgical instruments and to suture a prefabricated 4mm wide elastic strip under the microscope using Digital Surgicals MicroTrainer. The control group was taught continuously over 8hrs while the treatment group was taught in 2-hour sessions held each week over a span of 4 weeks. The learning outcomes that were measured included duration taken as well as the placement of the sutures in relation to each other, with the latter being objectively assessed with the use of a computer program from Digital Surgicals. In addition to being assessed at the beginning of the sessions, all participants completed another test 1 month after the completion of the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Medical students

Exclusion Criteria:

* Anyone who has been exposed to any form of microsurgical training

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Duration | For the mass learning group, at the end of the 1-day teaching session; for the spaced learning group, at the end of 1 month of teaching sessions.
  Duration taken to place pre-determined number of sutures on elastic strip
Suture density and alignment | For the mass learning group, at the end of the 1-day teaching session; for the spaced learning group, at the end of 1 month of teaching sessions.
  Another primary outcome measure is the objective scoring of the placement of sutures using a computer program from Digital Surgicals. In particular, the alignment and spacing of the sutures in relation to each other were assessed.

SECONDARY OUTCOMES:
Retention of skills - assessing duration | 1 month after the end of the final teaching session
  Duration taken to place pre-determined number of sutures on elastic strip - to assess retention of skills at 1 month after the completion of teaching sessions.
Retention of skills - assessing suture density and alignment | 1 month after the end of the final teaching session
  Assess retention of skills by assessing the suture density and alignment at 1 month after the completion of teaching sessions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjork RA: Retrieval practice and the maintenance of knowledge. In: Practical Aspects of Memory: Current Research and Issues. Edited by MM Gruneberg, PE Morris and RN Sykes. New York: John Wiley & Sons 1988; pp 396-401.
- [Background] Barsuk JH, Cohen ER, McGaghie WC, Wayne DB. Long-term retention of central venous catheter insertion skills after simulation-based mastery learning. Acad Med. 2010 Oct;85(10 Suppl):S9-12. doi: 10.1097/ACM.0b013e3181ed436c. PMID 20881713
- [Background] Boettcher M, Boettcher J, Mietzsch S, Krebs T, Bergholz R, Reinshagen K. The spaced learning concept significantly improves training for laparoscopic suturing: a pilot randomized controlled study. Surg Endosc. 2018 Jan;32(1):154-159. doi: 10.1007/s00464-017-5650-6. Epub 2017 Jun 22. PMID 28643052
- [Background] Brewster LP, Risucci DA, Joehl RJ, Littooy FN, Temeck BK, Blair PG, Sachdeva AK. Management of adverse surgical events: a structured education module for residents. Am J Surg. 2005 Nov;190(5):687-90. doi: 10.1016/j.amjsurg.2005.07.003. PMID 16226940
- [Background] Bridges M, Diamond DL. The financial impact of teaching surgical residents in the operating room. Am J Surg. 1999 Jan;177(1):28-32. doi: 10.1016/s0002-9610(98)00289-x. PMID 10037304
- [Background] Cecilio-Fernandes D, Cnossen F, Jaarsma DADC, Tio RA. Avoiding Surgical Skill Decay: A Systematic Review on the Spacing of Training Sessions. J Surg Educ. 2018 Mar-Apr;75(2):471-480. doi: 10.1016/j.jsurg.2017.08.002. Epub 2017 Aug 24. PMID 28843958
- [Background] Glenberg AM, Lehmann TS. Spacing repetitions over 1 week. Mem Cognit. 1980 Nov;8(6):528-38. doi: 10.3758/bf03213772. No abstract available. PMID 7219173
- [Background] Kerfoot BP, Fu Y, Baker H, Connelly D, Ritchey ML, Genega EM. Online spaced education generates transfer and improves long-term retention of diagnostic skills: a randomized controlled trial. J Am Coll Surg. 2010 Sep;211(3):331-337.e1. doi: 10.1016/j.jamcollsurg.2010.04.023. Epub 2010 Jul 13. PMID 20800189
- [Background] Kerfoot BP. Learning benefits of on-line spaced education persist for 2 years. J Urol. 2009 Jun;181(6):2671-3. doi: 10.1016/j.juro.2009.02.024. Epub 2009 Apr 16. PMID 19375095
- [Background] Lahiri A, Sebastin SJ, Yusoff SK, Sze Chong AK. Computer Aided Assessment in Microsurgical Training. J Hand Surg Asian Pac Vol. 2016 Jun;21(2):212-21. doi: 10.1142/S2424835516500211. PMID 27454636
- [Background] McGaghie WC, Issenberg SB, Petrusa ER, Scalese RJ. A critical review of simulation-based medical education research: 2003-2009. Med Educ. 2010 Jan;44(1):50-63. doi: 10.1111/j.1365-2923.2009.03547.x. PMID 20078756
- [Background] Moulton CA, Dubrowski A, Macrae H, Graham B, Grober E, Reznick R. Teaching surgical skills: what kind of practice makes perfect?: a randomized, controlled trial. Ann Surg. 2006 Sep;244(3):400-9. doi: 10.1097/01.sla.0000234808.85789.6a. PMID 16926566
- [Background] Pashler H, Rohrer D, Cepeda NJ, Carpenter SK. Enhancing learning and retarding forgetting: choices and consequences. Psychon Bull Rev. 2007 Apr;14(2):187-93. doi: 10.3758/bf03194050. PMID 17694899
- [Background] Patocka C, Khan F, Dubrovsky AS, Brody D, Bank I, Bhanji F. Pediatric resuscitation training-instruction all at once or spaced over time? Resuscitation. 2015 Mar;88:6-11. doi: 10.1016/j.resuscitation.2014.12.003. Epub 2014 Dec 13. PMID 25511519
- [Background] Spruit EN, Band GP, Hamming JF. Increasing efficiency of surgical training: effects of spacing practice on skill acquisition and retention in laparoscopy training. Surg Endosc. 2015 Aug;29(8):2235-43. doi: 10.1007/s00464-014-3931-x. Epub 2014 Oct 16. PMID 25318372
- [Background] Wojcik BM, Fong ZV, Patel MS, Chang DC, Petrusa E, Mullen JT, Phitayakorn R. The Resident-Run Minor Surgery Clinic: A Pilot Study to Safely Increase Operative Autonomy. J Surg Educ. 2016 Nov-Dec;73(6):e142-e149. doi: 10.1016/j.jsurg.2016.08.016. PMID 27886972
- [Background] Ziv A, Erez D, Munz Y, Vardi A, Barsuk D, Levine I, Benita S, Rubin O, Berkenstadt H. The Israel Center for Medical Simulation: a paradigm for cultural change in medical education. Acad Med. 2006 Dec;81(12):1091-7. doi: 10.1097/01.ACM.0000246756.55626.1b. PMID 17122476